CLINICAL TRIAL: NCT04258540
Title: The Effects of Yoga on Student Mental Health: A Randomised Controlled Trial
Brief Title: The Effects of Yoga on Student Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Tiril Elstad, Principal Investigator, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016/1751 C
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Mental Health; Public Health; Depression, Anxiety; Sleep Problem; University Students
Keywords: mental health; public health; depression; anxiety; sleep problems; insomnia; yoga; students
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders; Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomisation by a simple online program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group received a yoga course for 12 weeks, two times a week. Each yoga class was 1.25 hr in duration.
  Interventions: Behavioral: Yoga group
- Control group waitlist (Active Comparator): The control group were on a waitlist during the period of measurements, and received the same yoga course after all measurements had been completed.
  Interventions: Behavioral: yoga course

INTERVENTIONS:
Behavioral: Yoga group — The intervention group received yoga 2 times a week for 12 weeks (á 1.25 hr).
  Other Names: Intervention group
  Arms: Intervention group
Behavioral: yoga course — yoga course
  Arms: Control group waitlist

SUMMARY:
The investigators performed a randomised controlled trial with 202 healthy university students in the Oslo area, with 50:50 in a yoga intervention group and a waitlist control group. Measures included symptoms of depression and anxiety, sleep problems, heart rate variability (HRV), well-being and mindfulness at week 0 (baseline), week 12 (post-intervention) and week 24 (follow-up).

DETAILED DESCRIPTION:
Universities around the world are facing an epidemic of mental health problems among their students. The problem is truly a public health issue, affecting many and with serious consequences. Moreover, the global burden of disease-agenda calls for effective interventions with lasting effects that have the potential to improve the mental health of young adults. In this study the investigators aimed to determine whether yoga, a popular and widely available mind-body practice, can improve student mental health.

The participants were randomly assigned to a yoga group or waitlist control group in a 1:1 ratio by a simple online randomisation program. The intervention group was offered 24 yoga sessions over 12 weeks. Measurements were taken at week 0 (baseline), week 12 (post-intervention), and week 24 (follow-up). The primary outcome was psychological distress assessed by the HSCL-25 questionnaire. Analysis was performed based on the intention to treat-principle.

The methods were laid out in a protocol, previously published on the website of the study. (available at http://yogastudy.tilda.ws/). The planned analyses were very straightforward and included a description of the study participants, and simple analyses of each of the a priori selected outcome measures. We have not included or excluded any variables post-hoc.

ELIGIBILITY:
Inclusion Criteria:

* Living in the Oslo area

Exclusion Criteria:

* No serious mental health diagnoses
* No recent major life crisis
* No systematic yoga practice during the prior six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Change in Psychological Distress | Week 0 (baseline), week 12 (post-intervention) and week 24 (follow-up)
  Measured with the Hopkins Symptom Checklist 25 (HSCL-25) questionnaire. Consists of 25 items on symptoms of depression and anxiety, each rated on a 1 (not at all) to 4 (very much) scale. Total scores range from 1 to 4, a higher score indicating more psychological distress.

SECONDARY OUTCOMES:
Change in Heart Rate Variability (HRV) | Week 0 (baseline) and week 12 (post-intervention)
  Measured with nocturnal RMSSD (root mean square of successive differences), which is a validated measure of activity in the parasympathetic part of the autonomic nervous system. In general, an increase in RMSSD is associated with increased parasympathetic system activity and less distress.
Change in Mental Well-being | Week 0 (baseline), week 12 (post-intervention) and week 24 (follow-up).
  Measured with the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS), a 14-item Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). This scale has five response categories (from "not at all" to "all the time") that are added together to produce a total score ranging from 14 to 70. Higher scores indicate higher levels of mental well-being.
Change in Life Satisfaction | week 0 (baseline), week 12 (post-intervention) and week 24 (follow-up).
  Measured with the Satisfaction With Life Scale (SWLS), a 5-item questionnaire. Items are scored on a 1- to 7-point Likert scale. The total score is computed by adding all response values (ranging from 5 to 35), with higher scores indicating higher satisfaction.
Change in Mindfulness | Week 0 (baseline), week 12 (post-intervention) and week 24 (follow-up).
  Mindful Attention Awareness Scale, MAAS, a 15-item scale. The total score was computed by adding the score value on all individual items, producing a total score ranging from 15 to 75, with higher scores indicating higher levels of mindfulness.
Change in Sleep Problems | Week 0 (baseline), week 12 (post-intervention) and week 24 (follow-up).
  The investigators used the Bergen Insomnia Scale (BIS), a 6-item scale. Scores from 0 (no bad nights during the course of a week) to 7 (all nights) give a total score ranging from 0 to 42 (higher scores indicating more troubled sleep and daytime tiredness).

CONTACTS AND LOCATIONS:
Overall Officials: Tiril Elstad, MA (hon), Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elstad T, Ulleberg P, Klonteig S, Hisdal J, Dyrdal GM, Bjorndal A. The effects of yoga on student mental health: a randomised controlled trial. Health Psychol Behav Med. 2020 Nov 11;8(1):573-586. doi: 10.1080/21642850.2020.1843466. PMID 34040886